CLINICAL TRIAL: NCT00901199
Title: Safety of Deferasirox (ICL670) and Deferoxamine (Desferal or DFO) Combined Chelation Therapy in Patients With Transfusion Dependent Thalassemia and Iron Overload
Brief Title: Combined Chelation Therapy in Patients With Transfusion Dependent Thalassemia and Iron Overload
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elliott Vichinsky (Other)
Responsible Party: Sponsor-Investigator, Elliott Vichinsky, Director, Hematology/Oncology, UCSF Benioff Children's Hospital Oakland
Organization: UCSF Benioff Children's Hospital Oakland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AUS24T
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Thalassemia; Iron Overload
Keywords: Thalassemia; Chelation; Iron Overload; Thalassemia patients with Iron overload
MeSH Terms: conditions — Thalassemia; Iron Overload | interventions — Deferasirox; Deferoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deferasirox (Exjade) and Deferoxamine (DFO) (Experimental): All subjects received Deferasirox (Exjade) and Deferoxamine (DFO) dosing based on the iron overload at baseline.
  Interventions: Drug: Combo Chelation with Deferasirox (Exjade) and Deferoxamine (DFO)

INTERVENTIONS:
Drug: Combo Chelation with Deferasirox (Exjade) and Deferoxamine (DFO) — All subjects will be given Deferasirox 20-30 mg/kg for 7 days per week. All subject will be given Deferoxamine 50 mg/kg for 3-7 days per week. The number of days for Deferoxamine will be determined by liver iron concentration at baseline.
  Other Names: Deferasirox, (Exjade); Deferoxamine (DFO)

SUMMARY:
This is a pilot study looking at the safety and efficacy of giving combination chelation with deferasirox and deferoxamine. The hypothesis is that combination chelation is safe in decreasing overall iron in patients with thalassemia.

DETAILED DESCRIPTION:
This was a phase two pilot clinical trial designed to evaluate the safety and efficacy of the combination of deferasirox and deferoxamine in transfusion dependent thalassemia with a range of systemic iron burden. The duration of combined therapy was 12 months. Changes in liver iron concentration, ferritin, myocardial iron, and serum creatinine was monitored.

ELIGIBILITY:
Inclusion Criteria:

* Transfusion Dependent Thalassemia
* If iron between 5-15 mg/g dry liver by SQUID, subject must have a documented endocrinopathy or cardiac finding
* Older than 8 years

Exclusion Criteria:

* Participating on another interventional clinical trial

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Vichinsky, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- CHRCO, Oakland, California, United States

REFERENCES:
- [Result] Lal A, Porter J, Sweeters N, Ng V, Evans P, Neumayr L, Kurio G, Harmatz P, Vichinsky E. Combined chelation therapy with deferasirox and deferoxamine in thalassemia. Blood Cells Mol Dis. 2013 Feb;50(2):99-104. doi: 10.1016/j.bcmd.2012.10.006. Epub 2012 Nov 11. PMID 23151373

RESULTS

PARTICIPANT FLOW:
Groups:
- Deferasirox (Exjade) and Deferoxamine (DFO): Patients will receive combined chelation therapy using Deferasirox (Exjade) and Deferoxamine (DFO) with dosing based on liver iron concentration at baseline.
  Patients with moderate iron overload,defined as liver iron concentration of 5-15mg/g plus a documented endocrinopathy or cardiac iron (low MRI T2*), will receive 7 days per week of Deferasirox (Exjade) 20-30 mg/kg and Deferoxamine (DFO) 50 mg/kg 3-5 days per week.
  Patients with high iron overload, defined as liver iron concentration over 15mg/g will receive Deferasirox (Exjade) 20-30 mg/kg 7 days per week and Deferoxamine (DFO) 50 mg/kg 5-7 days per week.
Period: Overall Study
Arm/Group | Deferasirox (Exjade) and Deferoxamine (DFO)
Started | 22
Completed | 18
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Deferasirox (Exjade) and Deferoxamine (DFO)
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  Age, Categorical: <=18 years | 6
  Age, Categorical: Between 18 and 65 years | 16
  Age, Categorical: >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender Not Collected | 22

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Combined Treatment With Deferasirox and Deferoxamine Over 12 Months
Description: Change in liver iron concentration from baseline to 12 months with the use of combined chelation therapy. The change was calculated as the liver iron concentration at 12 months minus the value at baseline.
Time Frame: 12 months
Population: Eighteen subjects completed one year of therapy. Four subjects did not complete the study for the following reasons: lost to follow-up (1), abdominal pain (1), death (1), and non-compliance (1).
Measure: Median (Full Range); unit: mg/g
Groups:
- Deferasirox (Exjade) and Desferal (DFO): Subjects were treated with Deferasirox (Exjade) and Desferal (DFO) with dosing based on baseline iron overload.
Arm/Group | Deferasirox (Exjade) and Desferal (DFO)
Number analyzed (Participants) | 18
mg/g | -6.2 [-23.1 to 2.7]

2. Primary Outcome: Change in Serum Creatinine During 12 Months Combined Chelation Therapy
Description: Comparison of average serum creatinine over 12 months of combined chelation therapy compared with baseline serum creatinine.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Deferasirox (Exjade) and Desferal (DFO)
Number analyzed (Participants) | 22
mg/dl | 0.09 [0.05 to 0.12]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Deferasirox (Exjade) and Deferoxamine (DFO): Treatment with Deferasirox (Exjade) and Deferoxamine (DFO) with dosing based on baseline iron overload.
Arm/Group | Deferasirox (Exjade) and Deferoxamine (DFO)
All-Cause Mortality (participants affected / at risk) | 1/22
Serious Adverse Events (participants affected / at risk) | 2/22
Other Adverse Events (participants affected / at risk) | 1/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferasirox (Exjade) and Deferoxamine (DFO) (N=22)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) — Cholecystectomy
Central venous line infection (Infections and infestations) | 1 (1)
Death (Cardiac disorders) | 1 (1) — Baseline liver iron 24.6 mg/g, cardiac MRI T2* 4.8 ms, ejection fraction 67%. Two months into the study, presented to ER with abdominal pain, ascites, diarrhea, and leukocytosis. Expired during emergency colectomy from cardiac arrhythmias
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferasirox (Exjade) and Deferoxamine (DFO) (N=22)
Transfusion reaction (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No